CLINICAL TRIAL: NCT06549946
Title: A Phase I/II Open-label, Clinical Trial of Intratumoural Ixovex-1 as Single Agent Therapy or in Combination With Pembrolizumab in Palpable Solid Tumours
Brief Title: Ixovex-1 Single Agent and Combination Therapy
Acronym: IXACT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Psivac Ltd (Industry)
Collaborators: IQVIA Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ixovex-1-01
Record Dates: First submitted 2024-07-30; First posted 2024-08-12 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumor; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Open-label, single agent therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase Ia (Experimental): In Phase Ia, subjects will receive Ixovex-1 intratumourally.
  Interventions: Biological: Ixovex-1
- Phase Ib (Experimental): In Phase Ib, subjects will receive combination therapy with Ixovex-1 intratumourally and Pembrolizumab at the standard dose.
  Interventions: Biological: Ixovex-1; Biological: Pembrolizumab
- Phase II (Experimental): In Phase II, subjects will receive combination therapy with Ixovex-1 intratumourally and Pembrolizumab at the standard dose.
  Interventions: Biological: Ixovex-1; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Ixovex-1 — Ixovex-1 is a novel oncolytic human adenovirus serotype 5.
Biological: Pembrolizumab — Humanised antibody
  Other Names: Keytruda
  Arms: Phase II; Phase Ib

SUMMARY:
This is an open-label, dose de-escalating, non-randomised, multi-centre phase I/II study to determine safety and efficacy of the oncolytic virus, Ixovex-1 administered by intratumoural (IT) injection. This will be assessed in patients with palpable locally advanced, unresectable, or metastatic tumours, for whom all approved therapeutic options have been exhausted, are not available, are unlikely to have significant clinical benefit, or are declined by the patient.

DETAILED DESCRIPTION:
The Phase Ia arm of the study will employ a modified 3+3 dose de-escalation design. At least six subjects will receive intratumoural injections of Ixovex-1 approximately every 2 weeks over a period of 8 weeks (4 treatments) to determine the maximum tolerated dose (MTD).

The Phase Ib arm of the study will also employ a modified 3+3 dose de-escalation design. At least six subjects will be treated with Ixovex-1 (MTD from Phase Ia) in combination with standard dosing of Pembrolizumab to determine the recommended phase 2 dose (RP2D) for the combination therapy. Subjects will receive a total of 4 doses of Ixovex-1 and 8 doses of Pembrolizumab. Two treatments of Ixovex-1 will be given prior to commencing Pembrolizumab, and 2 treatments will be given in combination with the first 2 Pembrolizumab standard infusions administered every 3 weeks. The subsequent 6 doses of Pembrolizumab will be administered without Ixovex-1 every 3 weeks thereafter.

The Phase II arm of the study will use a Simon Type II study design to assess the RP2D of Ixovex-1 in combination with Pembrolizumab, as determined in Phase Ib. This will initially involve 6 subjects, with the potential to expand to 18 subjects in specific tumor types where clinical benefit or a positive treatment response is observed, such as in subjects who have previously been refractory to immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Have signed an informed consent indicating that the subject is aware of the neoplastic nature of their disease and have been informed of the procedures of the protocol, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts.
2. Female or male subjects aged ≥18 years (local regulatory requirements should be followed if the legal age of consent for study participation is >18 years old).
3. Subjects with injectable locally advanced, unresectable, or metastatic solid tumours.
4. In Phase Ia and Phase Ib, all solid tumour types will be accepted.
5. For Phase II, all solid tumour types will be considered with an emphasis on cutaneous squamous cell cancers and head and neck cancers.
6. Subjects with at least 1 measurable tumour (per RECIST 1.1) cutaneous/subcutaneous/nodal tumour suitable for direct percutaneous injection. Subjects may have other sites of disease.
7. A minimum of one tumour with a diameter of greater than 1 cm as measured by ultrasound and/or clinical measurement.
8. All approved therapeutic options have been exhausted, are not available, are unlikely to have significant clinical benefit or have been declined by the subject.
9. The Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
10. Life expectancy more than 6 months.
11. Pathologically documented, locally advanced, or metastatic solid malignancy.
12. Subject having laboratory values defined as:

    1. White blood cell counts greater than 3,000/mm3 OR absolute neutrophil counts greater than 1,500/mm3;
    2. Platelet count greater than 100,000/mm3;
    3. Haemoglobin greater than 9 g/dL (transfusions allowed if not used solely to meet eligibility criteria);
    4. Aspartate aminotransferase/alanine aminotransferase less than 2.5 times ULN;
    5. Bilirubin no greater than 1.5 times ULN;
    6. Creatinine clearance (Cockcroft-Gault formula) ≥50 mL/min.
13. Be willing and able to comply with scheduled visits, the treatment plan, imaging, and laboratory tests.

Exclusion Criteria:

1. Presence of overt leptomeningeal or active central nervous system (CNS) metastases, or CNS metastases that require local CNS-directed therapy (eg, radiotherapy or surgery) or increasing doses of corticosteroids within the prior 2 weeks. Subjects with treated brain metastases should be neurologically stable (for 4 weeks post treatment and prior to study enrolment) and off steroids for at least 2 weeks before administration of any study treatment.
2. Tumours involving a major blood vessel where tumour necrosis might endanger the subject.
3. Impaired cardiac function or clinically significant cardiac disease, including any of the following:

   1. Clinically significant and/or uncontrolled heart disease such as congestive heart failure requiring treatment (New York Heart Association Grade ≥2), left ventricular ejection fraction <50% as determined by multiple gated acquisition (MUGA) or echocardiogram (ECHO), uncontrolled hypertension, or clinically significant arrhythmia.
   2. Acute myocardial infarction or unstable angina pectoris <6 months prior to study entry.
4. Subjects with interstitial pneumonia or history of drug-induced interstitial pneumonia/pneumonitis.
5. Have an immune system disorder (known human immunodeficiency virus infection or hepatitis B or C).
6. Chronic liver disease or chronic hepatitis (Child-Pugh class B or C hepatic impairment).
7. Malignant disease, other than that being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to study treatment; completely resected basal cell and squamous cell skin cancers; any malignancy considered to be indolent and that has never required therapy; and completely resected carcinoma in situ of any type.
8. Subjects receiving systemic chronic steroid therapy or any immunosuppressive therapy (>10 mg/day prednisone or equivalent). Topical, inhaled, nasal, and ophthalmic steroids are allowed.
9. Use of any live vaccines against infectious diseases within 4 weeks of initiation of study treatment.
10. Subjects with a history of stroke or having active neurological symptoms, with the exception of chronic conditions which, in the opinion of the neurologist, Investigator, and the Sponsor, would not impact ongoing neurologic assessments while on study treatment.
11. Active infection requiring systemic or antiviral or antibiotic therapy.
12. Subjects with active cytomegalovirus infection.
13. Prior therapy:

    1. Major surgery within 2 weeks of the first dose of study treatment (mediastinoscopy, insertion of a central venous access device, and insertion of a feeding tube are not considered major surgery).
    2. Did not recover from prior biologic therapy, endocrine therapy, or any prior diagnostic or therapeutic procedures.
    3. Received prior chemotherapy within 21 days of C1D1.
    4. Previous treatment with oncolytic virotherapy.
14. Presence of CTCAE ≥ Grade 2 toxicity (except alopecia, peripheral neuropathy, and ototoxicity, which are excluded if ≥ CTCAE Grade 3) due to prior cancer therapy.
15. Participation in an interventional, investigational study within 4 weeks or 5 half-lives (whichever is shorter) of the first dose of study treatment.
16. Any medical condition that would, in the Investigator's judgement, prevent the subject's participation in the clinical study due to safety concerns, compliance with clinical study procedures, or interpretation of study results.
17. Pregnant or breastfeeding woman (pregnant or lactating women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin laboratory test). Female subjects of childbearing potential must agree to use highly effective contraception (during the study and for 6 months from last dose of Ixovex-1), must be surgically sterile, or must be postmenopausal. Male subjects must use a condom (during the study and for 6 months from last dose of Ixovex-1) or be surgically sterile. Additionally, female partners may be requested to use highly effective contraception as an additional safeguard. For Pembrolizumab, the manufacturer recommends contraception for women of childbearing age during treatment with Pembrolizumab and for 4 months post last treatment of Pembrolizumab. For Pembrolizumab, the manufacturer recommends contraception for male subjects during treatment with Pembrolizumab and for 4 months post last treatment of Pembrolizumab.
18. Known hypersensitivity to any component of Ixovex-1 or pembrolizumab (latter for Phase 1b and Phase 2 only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
To determine the safety profile of Ixovex-1 when administered by intratumoural injection alone or in combination with Pembrolizumab in patients with unresectable, locally advanced, or metastatic solid tumours. | Through study completion, an average of 2 years
  Percentage of subjects with DLTs during the DLT period [Day 1 to Day 28].
  Percentage of subjects with SAEs, overall and by maximum severity [Day 1 to 30 days after last dose].
  Percentage of subjects with TEAEs, overall and by maximum severity [Day 1 to 30 days after last dose].
To determine the MTD and recommended Phase 2 dose of Ixovex-1. | Through study completion, an average of 2 years
  Percentage of subjects with TEAEs, overall and by maximum severity [Day 1 to 30 days after last dose].

SECONDARY OUTCOMES:
To assess clinical efficacy using a combination of radiological imaging, medical photography, and histology. | Through study completion, an average of 2 years
  Overall response rate (CR + PR).
  Best overall confirmed response - percentage of subjects at each response level (CR, PR, SD, PD).
Assessment of antitumour effects in injected tumours and in non-injected tumours. | Through study completion, an average of 2 years
  Change in cumulative tumour size.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Harrington, Principal Investigator — The Royal Marsden
Locations (1):
- The Royal Marsden, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anwar M, Arendt ML, Ramachandran M, Carlsson A, Essand M, Akusjarvi G, Alusi G, Oberg D. Ixovex-1, a novel oncolytic E1B-mutated adenovirus. Cancer Gene Ther. 2022 Nov;29(11):1628-1635. doi: 10.1038/s41417-022-00480-3. Epub 2022 May 20. PMID 35596069